CLINICAL TRIAL: NCT04678518
Title: Inflammatory Markers Dynamics in Response to Extra-corporeal Membrane Oxygenator Decannulation
Acronym: ECMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: MRC-01-20-155
Record Dates: First submitted 2020-10-20; First posted 2020-12-22 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Markers Changes in Response to Extra-corporeal Membrane Oxygenator Decannulation

STUDY DESIGN:
Intervention Model Description: The study will be conducted in the Heart Hospital to be conducted from the time of ethical approval for 24 months.
  The clinical characterization of post decannulation SIRS when patient fulfill 2 out of 3 criteria, fever (temperature >38.3 Celsius), leukocytosis (white blood cell [WBC] >12,000, or > 25% increase from pre-procedure baseline), and need for escalation of vasopressors post decannulation. The rest of SIRS criteria will not be used as it is subjected to changes due to contribution from the inotropes, sedation, pain level and ventilation settings. [12] Patients will be grouped according to the presence or absence of SIRS criteria into group I (SIRS) and group II (no-SIRS). Inflammatory makers that will include Interleukins (IL); IL1, IL2, IL6 and TNF 1 hour before decannulation and 3 times after decannulation (1 hours, 12 hours and 24 hours) both groups will be compared.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIRS (Active Comparator): Patients will be grouped according to the presence or absence of SIRS criteria into group I (SIRS)
  Interventions: Diagnostic Test: Inflammatory makers that will include Interleukins (IL); IL1, IL2, IL6 and TNF
- NON-SIRS (Placebo Comparator): Patients will be grouped according to the presence or absence of SIRS criteria into group II (Non-SIRS)
  Interventions: Diagnostic Test: Inflammatory makers that will include Interleukins (IL); IL1, IL2, IL6 and TNF

INTERVENTIONS:
Diagnostic Test: Inflammatory makers that will include Interleukins (IL); IL1, IL2, IL6 and TNF — 1 hour before decannulation and 3 times after decannulation (1 hours, 12 hours and 24 hours)

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) aim at providing cardiac, respiratory support, or both. The use of ECMO could be associated with systemic inflammatory response syndrome (SIRS) at the time of initiation or the time of decannulation. There is an existing evidence to state that clinical criteria of SIRS accompany decannulation. We aim at proving this relation through studying the inflammatory markers changes before and after decannulation. The investigators will study all participants who require ECMO support in the heart hospital, all patient will be subjected to clinical evaluation of the SIRS criteria plus studying the inflammatory makers that will include IL1, IL2, IL6 and TNF before and after decannulation. Participants will be divided based on the SIRS criteria into 2 groups and both groups will be compared using Chi-Square analysis (Fisher tests if small sample size) or two tailed t-test, as appropriate

ELIGIBILITY:
Inclusion Criteria:

* ALL ECMO patients candidates for decannulation

Exclusion Criteria:

* patients who have identified sepsis prior to decannulation, febrile patients, patient who receive steroids and patient who die within 48 hours after ECMO decannulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine changes | 2 years
  Cytokines changes: Interleukins (IL); IL1, IL2, IL6 and TNF 1 hour before decannulation and 3 times after decannulation (1 hours, 12 hours and 24 hours)

OTHER OUTCOMES:
Length of stay in ICU | First 48 hours after ECMO initiation
Length of mechanical ventilation | First 48 hours after ECMO initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad medical corporation, Doha, DA, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hill JD, O'Brien TG, Murray JJ, Dontigny L, Bramson ML, Osborn JJ, Gerbode F. Prolonged extracorporeal oxygenation for acute post-traumatic respiratory failure (shock-lung syndrome). Use of the Bramson membrane lung. N Engl J Med. 1972 Mar 23;286(12):629-34. doi: 10.1056/NEJM197203232861204. No abstract available. PMID 5060491
- [Result] Sauer CM, Yuh DD, Bonde P. Extracorporeal membrane oxygenation use has increased by 433% in adults in the United States from 2006 to 2011. ASAIO J. 2015 Jan-Feb;61(1):31-6. doi: 10.1097/MAT.0000000000000160. PMID 25303799
- [Result] Davies MG, Hagen PO. Systemic inflammatory response syndrome. Br J Surg. 1997 Jul;84(7):920-35. doi: 10.1002/bjs.1800840707. PMID 9240130
- [Result] Wang S, Krawiec C, Patel S, Kunselman AR, Song J, Lei F, Baer LD, Undar A. Laboratory Evaluation of Hemolysis and Systemic Inflammatory Response in Neonatal Nonpulsatile and Pulsatile Extracorporeal Life Support Systems. Artif Organs. 2015 Sep;39(9):774-81. doi: 10.1111/aor.12466. Epub 2015 May 1. PMID 25940752
- [Result] Rungatscher A, Tessari M, Stranieri C, Solani E, Linardi D, Milani E, Montresor A, Merigo F, Salvetti B, Menon T, Faggian G. Oxygenator Is the Main Responsible for Leukocyte Activation in Experimental Model of Extracorporeal Circulation: A Cautionary Tale. Mediators Inflamm. 2015;2015:484979. doi: 10.1155/2015/484979. Epub 2015 May 4. PMID 26063972
- [Result] McILwain RB, Timpa JG, Kurundkar AR, Holt DW, Kelly DR, Hartman YE, Neel ML, Karnatak RK, Schelonka RL, Anantharamaiah GM, Killingsworth CR, Maheshwari A. Plasma concentrations of inflammatory cytokines rise rapidly during ECMO-related SIRS due to the release of preformed stores in the intestine. Lab Invest. 2010 Jan;90(1):128-39. doi: 10.1038/labinvest.2009.119. Epub 2009 Nov 9. PMID 19901912
- [Result] Graulich J, Walzog B, Marcinkowski M, Bauer K, Kossel H, Fuhrmann G, Buhrer C, Gaehtgens P, Versmold HT. Leukocyte and endothelial activation in a laboratory model of extracorporeal membrane oxygenation (ECMO). Pediatr Res. 2000 Nov;48(5):679-84. doi: 10.1203/00006450-200011000-00021. PMID 11044491
- [Result] Shi J, Chen Q, Yu W, Shen J, Gong J, He C, Hu Y, Zhang J, Gao T, Xi F, Li J. Continuous renal replacement therapy reduces the systemic and pulmonary inflammation induced by venovenous extracorporeal membrane oxygenation in a porcine model. Artif Organs. 2014 Mar;38(3):215-23. doi: 10.1111/aor.12154. Epub 2013 Dec 11. PMID 24329567
- [Result] Yimin H, Wenkui Y, Jialiang S, Qiyi C, Juanhong S, Zhiliang L, Changsheng H, Ning L, Jieshou L. Effects of continuous renal replacement therapy on renal inflammatory cytokines during extracorporeal membrane oxygenation in a porcine model. J Cardiothorac Surg. 2013 Apr 29;8:113. doi: 10.1186/1749-8090-8-113. PMID 23628149
- [Result] Warren OJ, Watret AL, de Wit KL, Alexiou C, Vincent C, Darzi AW, Athanasiou T. The inflammatory response to cardiopulmonary bypass: part 2--anti-inflammatory therapeutic strategies. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):384-93. doi: 10.1053/j.jvca.2008.09.007. Epub 2008 Dec 3. No abstract available. PMID 19054695
- [Result] Thangappan K, Cavarocchi NC, Baram M, Thoma B, Hirose H. Systemic inflammatory response syndrome (SIRS) after extracorporeal membrane oxygenation (ECMO): Incidence, risks and survivals. Heart Lung. 2016 Sep-Oct;45(5):449-53. doi: 10.1016/j.hrtlng.2016.06.004. Epub 2016 Jul 15. PMID 27425197
- [Result] Lamb KM, Hirose H, Cavarocchi NC. Preparation and technical considerations for percutaneous cannulation for veno-arterial extracorporeal membrane oxygenation. J Card Surg. 2013 Mar;28(2):190-2. doi: 10.1111/jocs.12058. Epub 2013 Feb 5. PMID 23379727
- [Result] Shaheen A, Tanaka D, Cavarocchi NC, Hirose H. Veno-Venous Extracorporeal Membrane Oxygenation (V V ECMO): Indications, Preprocedural Considerations, and Technique. J Card Surg. 2016 Apr;31(4):248-52. doi: 10.1111/jocs.12690. Epub 2016 Feb 3. PMID 26842109
- [Derived] Bilal O, Omar AS, Tbishat L, Salama A, Prabhu KS, Uddin S, Kaddoura R, Carr CS, Taha R, Pattath A, Alkhulaifi A. Pro-inflammatory cytokines in response to systemic inflammatory response syndrome post extra-corporeal membrane oxygenator decannulation. Int J Artif Organs. 2026 Jan;49(1):30-38. doi: 10.1177/03913988251398846. Epub 2025 Dec 11. PMID 41383076